CLINICAL TRIAL: NCT01125982
Title: Postanaesthetic Outcome and Assessment of Fatigue in Day-surgery Laparoscopic Cholecystectomy
Brief Title: Postoperative Fatigue and Nausea Related to Choice of Anaesthetic Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Torkjell Nostdahl, MD, Anaesthesiologist, Sykehuset Telemark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009/2171(REK); 2009-017117-30 (EudraCT Number); 09/15863 (Other: Norwegian Medicines Agency)
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Fatigue; Nausea
MeSH Terms: conditions — Fatigue; Nausea | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): Patients will receive Desflurane to provide sleep during anaesthesia for laparoscopic cholecystectomy. Analgesia will be provided by remifentanil.
  Interventions: Drug: Desflurane
- Propofol (Active Comparator): Patients will receive Propofol to provide sleep during anaesthesia for laparoscopic cholecystectomy. Analgesia will be provided by remifentanil.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Continuous intravenous infusion at 3-6 µg/mL (Ce - Target Controlled Infusion) during anaesthesia to provide sleep.
  Arms: Propofol
Drug: Desflurane — Continuous inhalation at 0.7-0.8 MAC (endtidal) during anaesthesia to provide sleep
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
The purpose of this study is to establish validated outcome measures for Postoperative Fatigue and Postoperative nausea, and to compare clinical impact of postanaesthetic symptoms during first week after Propofol or Desflurane based anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for day-surgery laparoscopic cholecystectomy
* The patient is able to read and comprehend Norwegian language
* The patient is cognitive adequate and able to fill in survey forms
* The patient has read and signed patient information form

Exclusion Criteria:

* Serious illness (ASA 3-4)
* Pregnancy or suspected pregnancy
* Breastfeeding women
* Contraindications to use of NSAIDs
* Serious allergic reaction to anaesthetics
* Allergy towards egg, soya or peanuts
* Known or suspected Malignant Hyperthermia or Porphyria
* Fatigue-related diagnosis
* Recently received adjuvant therapy (chemotherapy, radiotherapy)
* Severe chronic pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of fatigue after anaesthesia based on propofol or desflurane | Within the first week postoperatively
  Fatigue scales; Chalder Fatigue Scale and Incidence-Consequence Fatigue Scale. Measure points; 1st, 3rd, 6th and 30th day postoperatively.

SECONDARY OUTCOMES:
Incidence and severity of postoperative nausea after anaesthesia based on propofol or desflurane | Within the first week postoperatively
  PONV scales; 4-point Likert Scale and 11-point NRS Scale.
  Measure points; 1st, 3rd, 6th and 30th day postoperatively.
Fatigue scale validation | See under "Description":
  To ensure validated outcome measures we will perform validation and comparison of two different fatigue scales (Chalder Fatigue Scale and Identity-Consequences Fatigue Scale). This will primarily be performed in a mixed surgical population. In addition the scales will also be validated in palliative patients, patients with possible CFS/ME diagnosis and patients with chronic pain.
  Data aquisition will be cross-sectional, but the surgical population will also yield longitudinal data (preop. and 3rd postoperative day)

CONTACTS AND LOCATIONS:
Locations (1):
- Telemark Hospital, Skien, Telemark, Norway